CLINICAL TRIAL: NCT01454336
Title: Phase 1 Trial of Combined Pioglitazone Plus Autologous Bone Marrow Mesenchymal Stem Cell Transplantation in Patients With Compensated Cirrhosis
Brief Title: Transplantation of Autologous Mesenchymal Stem Cell in Decompensate Cirrhotic Patients With Pioglitazone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-liver-003
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2010-02

CONDITIONS: Liver Fibrosis
Keywords: MSCs; Pioglitazon; fibrosis; liver
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cirrhotic Patients (Experimental): 3 cirrhotic patients who underwent a combination of cell therapy and chemotherapy
  Interventions: Biological: Cell injection

INTERVENTIONS:
Biological: Cell injection — MSCs introduced into portal vein

SUMMARY:
Liver cirrhosis (LC) is the final destiny in chronic liver disease. Liver transplantation is the only effective therapy available to these patients. However, limited number of donors, post surgical complications, immunological rejection, and financial considerations are it's essential problems. The immuomodulatory impact of MSCs in fibrosis was confirmed, and several clinical studies have applied MSCs to eliminate the progression of fibrosis. In this research the investigators will study the affect of MSCs and Pioglitazone in the process of fibrosis.

DETAILED DESCRIPTION:
BM Aspiration will be done twice (6 months interval) from the iliac crest according to standard procedures under general anesthesia and is collected (200ML) in plastic bags containing anti coagulant. After precipitation of red blood cells, mononuclear cells will be collected by centrifugation in Ficoll-Paque density gradient. MNCs will be cultured in T150 flasks. Cells will be expanded in several subcultures.MSCs will be injected (6 months interval) via portal vein under sonography monitoring.Each patient will receive 30mg Pioglitazone daily for 24 months. After cell therapy, patients are followed up every week for 6 months, and laboratory data are analyzed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 Years cirrhotic patient
* Approved cirrhosis by elastografy ,biopsy, sonography

Exclusion Criteria:

1 - Portal vein thrombosis 2-Hepatic encephalopathy, score 3&4 3-ALT & AST 3times more than normal 4-Serum Cr more than 1/5mg/dL 5-(Anti-HIV +) (Anti-HCV+) (HBS-Ag+) 6-Hepatocel carcinoma 7- Primary sclerosing cholangitis (PSC) 8- Esophageal varices grade 4 9-Addiction 10-Child Score B,C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
ALT | 12 months
  Evaluation of ALT levels during 12 months
AST | 12 months
  Evaluation of AST levels after intervention during 12 months
Serum Albumin | 12 months
  The evaluation of serum albumin levels for 12 months
Liver Fibrosis | 12 months
  The decrease in grade of liver fibrosis

SECONDARY OUTCOMES:
Progression of fibrosis | 12 months
  Evaluation of fibrosis based on fibroscan and biopsy and scoring

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Reza malekzadeh, MD, Study Director — Director of DDRC; Massoud vosough, MD,PhD, Principal Investigator — Royan regenerative medicine
Locations (1):
- Royan Institute, Tehran, Iran